CLINICAL TRIAL: NCT00972439
Title: Evaluating the Effect of Oral Contraceptive Progestin Dose on Breast Epithelial Cell Proliferation
Brief Title: Oral Contraceptive (OC) Progestin Dose and Breast Proliferation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HS-07-00269
Record Dates: First submitted 2009-09-03; First posted 2009-09-07 (Estimated); Results first posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2017-12

CONDITIONS: Oral Contraceptive
Keywords: Oral Contraceptives; Breast Tissue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ortho-Novum® 1/35 (Active Comparator): Ortho-Novum® 1/35 is an oral contraceptive that contains more progestin.
  Interventions: Drug: Oral Contraceptive: Ortho-Novum® 1/35
- Ovcon Fe® (Active Comparator): Ovcon Fe® is an oral contraceptive that contains less progestin.
  Interventions: Drug: Oral Contraceptive: Ovcon Fe®

INTERVENTIONS:
Drug: Oral Contraceptive: Ortho-Novum® 1/35
  Arms: Ortho-Novum® 1/35
Drug: Oral Contraceptive: Ovcon Fe®
  Arms: Ovcon Fe®

SUMMARY:
The purpose of this research study is to gain a better understanding of the changes that may occur in the breast when a woman uses an oral contraceptive (birth control pill). Some research indicates that women who use birth control pills with lower amounts of progestin (a hormone in the birth control pill) may have lower breast cell growth than women who use birth control pills with a higher amount of progestin; this research will examine that in detail.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-34.
2. Premenopausal.
3. Currently taking or want to start oral contraceptives for contraception
4. Non-smoker.
5. Competent to give informed consent (as judged by the investigator).
6. Provided written informed consent.
7. Willingness to refrain from smoking and consumption of grapefruit or grapefruit juice during the study (grapefruit interferes with metabolism of exogenously administered OCs).

Exclusion Criteria:1.

1. Abnormal breast examination.
2. History or current therapeutic or prophylactic use of anticoagulants.
3. Known bleeding disorder or history of unexplained bleeding or bruising.
4. History of breast cancer or previous diagnostic breast biopsy.
5. Known allergy to local anesthetic.
6. Currently pregnant or pregnant within the previous 6 months.
7. Having any standard contra-indication to being prescribed OCs.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2007-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DeShawn Taylor, M.D., Principal Investigator — University of Southern California
Locations (1):
- Los Angeles County Hospital, Los Angeles, California, United States

REFERENCES:
- [Derived] Hovanessian-Larsen L, Taylor D, Hawes D, Spicer DV, Press MF, Wu AH, Pike MC, Pearce CL. Lowering oral contraceptive norethindrone dose increases estrogen and progesterone receptor levels with no reduction in proliferation of breast epithelium: a randomized trial. Contraception. 2012 Sep;86(3):238-43. doi: 10.1016/j.contraception.2011.12.015. Epub 2012 Feb 9. PMID 22325110

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: April 2008 - October 2008 Ob/gyn clinics
Period: Overall Study
Arm/Group | Ortho-Novum® 1/35 | Ovcon Fe®
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ortho-Novum® 1/35 | Ovcon Fe® | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 33
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (4.4) | 28.1 (4.8) | 26.8 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Breast Cell Proliferation Levels Between the Two Oral Contraceptive Dose Groups
Description: Percent of cells expressing staining for Ki67 will be examined in breast epithelial cells
Time Frame: 32 weeks
Population: Five of the breast biopsy specimens contained insufficient TDLU epithelial tissue for analysis and one of the remaining women was diagnosed with a follicular cyst on the day of the biopsy, leaving 27 evaluable women.
Measure: Mean (95% Confidence Interval); unit: Percent of cells staining for Ki67
Arm/Group | Ortho-Novum® 1/35 | Ovcon Fe®
Number analyzed (Participants) | 14 | 13
Percent of cells staining for Ki67 | 7.5 [3.8 to 14.6] | 12.4 [6.3 to 24.2]

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning day 1 of study and continued throughout the study until 30 days after the last dose.
Arm/Group | Ortho-Novum® 1/35 | Ovcon Fe®
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No